CLINICAL TRIAL: NCT03999723
Title: Combining Active and Passive DNA Hypomethylation: A Randomized, Placebo-Controlled Phase II Study of the Efficacy and Safety of Oral Vitamin C in Combination With Azacitidine in Patients With Higher-Risk MDS, CMML-2 or Low-Blast Count AML
Brief Title: Combining Active and Passive DNA Hypomethylation
Acronym: EVI-3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kirsten Grønbæk (Other)
Collaborators: Van Andel Institute - Stand Up To Cancer Epigenetics Dream Team (Unknown); Karolinska University Hospital (Other); Skane University Hospital (Other); Sahlgrenska University Hospital (Other); University of Southern California (Other); Imperial College London (Other); University of Copenhagen (Other); Zealand University Hospital (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Technical University of Denmark (Other); Aarhus University Hospital (Other); Uppsala University Hospital (Other)
Responsible Party: Sponsor-Investigator, Kirsten Grønbæk, Professor, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-18040929
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia
Keywords: Vitamin C; Ascorbic acid; Azacitidine; Hypomethylating agents; Randomized, Placebo-Controlled Trial
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: A multicentre, randomized, parallel-group, placebo-controlled, double-blind phase 2 study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind masking (Participant, Care Provider, Investigator, (some) Outcomes Assessors)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Oral vitamin C (ascorbic acid) will be given in a dose of 1000 mg daily (two capsules of 500 mg once daily) starting day 1 in the 1st azacitidine (AZA) cycle (D1/C1) and continuing until discontinuation of AZA or end of study, whichever occurs earlier.
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Placebo will be administered orally as two capsules once daily that look and taste identical to the capsules containing vitamin C. Treatment will start day 1 in the 1st azacitidine (AZA) cycle (D1/C1) and continuing until discontinuation of AZA or end of study, whichever occurs earlier. The content of the placebo capsules is glucose monohydrate, potato starch, gelatin, magnesium stearate and talc.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — Oral vitamin C (ascorbic acid) 1000 mg daily will be administered from day 1 in the 1st AZA cycle (D1/C1) and continued until discontinuation of AZA or EOS as combination treatment.
  Other Names: Ascorbic acid
  Arms: Vitamin C
Dietary Supplement: Placebo — Placebo capsules (two capsules once daily) will be administered from day 1 in the 1st AZA cycle (D1/C1) and continued until discontinuation of AZA or EOS.
  Arms: Placebo

SUMMARY:
This is a multicentre, randomized, parallel-group, placebo-controlled, double-blind phase 2 study of the efficacy and safety of oral vitamin C supplement in combination with azacitidine in patients with higher-risk MDS, CMML-2 or low-blast count AML. The primary purpose is to investigate if oral vitamin C supplementation to azacitidine, compared with azacitidine + placebo, can increase the effectiveness of epigenetic therapy in patients with higher-risk myeloid malignancies, who are not candidates for allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
EVI-3 is a phase 2 international, multicentre, randomized, parallel-group, placebo-controlled, double-blind study of the efficacy and safety of oral vitamin C supplement in combination with azacitidine (AZA) in patients with higher-risk myeloid malignancies with or without mutations in genes recurrently affected in myeloid malignancies. Treatment allocation is in 1:1 ratio (vitamin C vs. placebo) by block randomization stratified by clinical site. Study entry is staggered. Patients are randomized to either oral vitamin C 1000 mg daily or placebo from start of AZA treatment until end of study (EOS) or until AZA treatment is discontinued at the discretion of the treating physician, whichever occurs earlier. The accrual time is estimated to 48 months and 6 months follow-up, thus, maximum treatment duration will be approximately 54 months. A total of 196 patients is planned for enrollment.

Study visits are scheduled at baseline, after 1st AZA treatment cycle, after 6 AZA treatment cycles, and, if AZA treatment is continued, at EOS or end of AZA treatment. Evaluations at study visits include bone marrow investigation, peripheral blood tests, patient-reported outcome measures, adverse events and compliance. Bone marrow aspirate and peripheral blood will be collected for biobank at each study visit.

All patients will undergo follow-up once yearly from EOS. Follow-up will include information on duration of AZA therapy, survival and disease progression from myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) to acute myeloid leukemia (AML), if diagnosed following a clinical indication for a bone marrow test.

ELIGIBILITY:
Inclusion Criteria:

• Patients eligible for treatment with azacitidine with one of the following diagnoses according to World Health Organization 2016:

* MDS Higher-risk MDS according to the IPSS-R, i.e., intermediate- to very high-risk (IPSS-R score > 3)
* CMML CMML with 10-29 percent marrow blasts without myeloproliferative disorder
* AML AML with 20-30 percent blasts (low-blast count AML)

Note: Patients with therapy-related MDS are eligible if they have not received radiation or chemotherapy for six months.

Exclusion Criteria:

* Patient eligible for allogeneic stem cell transplantation
* Prior therapy with hypomethylating agents
* Any matter constituting an exclusion criterion for treatment with azacitidine
* Patient receiving other active cancer treatment, including investigational agents, with the exception of hydroxyurea for white blood cell (WBC) control, G-CSF, and low permanent doses of steroid (≤ 25 mg oral prednisolone per day) for inflammatory disorders
* Therapeutic radiation or chemotherapy within the past 6 months
* History of allergic reactions to ascorbic acid
* History of kidney or urinary tract stones requiring intervention within the past year
* Lack of ability to understand the information given, or lack of willingness to sign a written informed consent document
* Unwillingness to comply with the protocol
* Unwillingness to discontinue any and all use of vitamin C medication/supplementation including multivitamin at least 3 days (but preferably longer) prior to inclusion and baseline sampling
* Planned azacitidine treatment after allogeneic stem cell transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status ≥3
* Uncontrolled comorbidity including impaired hepatic function (total serum bilirubin >1.5 × upper limit of the normal range (ULN), serum alanine transaminase >3 × ULN, chronic hepatitis with decompensated cirrhosis), disabling psychiatric disease, severe neurologic disease, severe metabolic disease, or severe cardiac disease (NYHA class 3-4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 0-54 months
  Event-free survival in months in the group of patients receiving oral vitamin C + AZA (arm A) vs. the group of patients receiving placebo + AZA (arm B) calculated from the time of randomization to EOS. Event is defined as death, relapse, progression or lack of a response at 6 AZA cycles as defined by IWG 2006 (MDS and CMML) and ELN 2017 (AML) response criteria

SECONDARY OUTCOMES:
Adverse events and serious adverse events | 0-54 months
  Number and ratio of patients with adverse events in arm A vs. arm B assessed from the time of administration of intervention (day 1, AZA cycle 1 = D1/C1) to EOS. Total number of adverse events and serious adverse events and the number per year from D1/C1 to EOS in arm A vs. arm B. Number of patients discontinuing the intervention and discontinuation rate in arm A vs. arm B from D1/C1 to EOS
Overall survival | 0-54 months
  Overall survival in months in arm A vs. arm B calculated from the time of randomization to EOS
Overall response rate | 0-54 months
  Rate of overall response and rates of individual responses (as according to international consensus criteria), including best response, in arm A vs. arm B after 6 AZA cycles and at EOS
Patient-reported outcome (PRO) measures | 0-54 months
  Change in PRO measures including health-related quality of life scores (EORTC QLQ-C30 and Hematological Malignancy (HM)-PRO) from baseline to end of 1st AZA cycle, after 6 AZA cycles and EOS, if AZA treatment ongoing, respectively, in arm A vs. arm B. Numerical PRO scores after the 1st AZA cycle and after 6 AZA cycles (and EOS), respectively, in arm A vs. arm B
Variant allele frequency (VAF) of mutated clones | 0-54 months
  Change in VAF of mutated clones (in percentage points and in percentage) in bone marrow mononuclear cells from baseline to end of 6th AZA cycle and to end of treatment (if occurring before EOS) in arm A vs. arm B. Number and ratio of patients with appearance of new mutations between baseline and end of 6th AZA cycle (and end of treatment) in arm A vs. arm B. Total number of new mutations in arm A vs. arm B from baseline to end of 6th AZA cycle (and end of treatment)
Global 5-hydroxymethylcytosine (5-hmC)/5-methylcytosine (5-mC) | 0-54 months
  Change in global 5-hmC/5-mC in bone marrow CD34+ cells from baseline to end of 1st AZA cycle, end of 6th AZA cycle and end of treatment (if occurring before EOS), respectively, in arm A vs. arm B. Global 5-hmC/5-mC in bone marrow CD34+ cells at end of 1st AZA cycle and end of 6th AZA cycle (and end of treatment), respectively, in arm A vs. arm B
Site specific 5-hmC/5-mC | 0-54 months
  Change in 5-hmC/5-mC at specific loci at promoters/enhancers/long terminal repeats (LTRs) or at other regulatory genomic regions of tumor suppressors, oncogenes, genes involved in hematopoietic development or human endogenous retrovirus (HERV) in bone marrow CD34+ cells from baseline to end of 1st AZA cycle, end of 6th AZA cycle and end of treatment (if occurring before EOS), respectively, in arm A vs. arm B. Site specific 5-hmC/5-mC in bone marrow CD34+ cells at end of 1st AZA cycle and end of 6th AZA cycle (and end of treatment), respectively, in arm A vs. arm B
Gene expression | 0-54 months
  Change in expression of genes involved in viral defense pathways, cell differentiation and tumor suppression and oncogenes in bone marrow CD34+ cells from baseline end of 1st AZA cycle, end of 6th AZA cycle and end of treatment (if occurring before EOS), respectively, in arm A vs. arm B. Expression of genes involved in viral defense pathways, cell differentiation and tumor suppression in bone marrow CD34+ cells at end of 1st AZA cycle and end of 6th AZA cycle (and end of treatment), respectively, in arm A vs. arm B
mRNA expression of HERV and HERV specific T-cell responses | 0-54 months
  Change in levels of mRNA expression of HERV in bone marrow CD34+ cells and HERV specific T-cell responses from baseline to end of 1st AZA cycle, end of 6th AZA cycle and end of treatment (if occurring before EOS), respectively, in arm A vs. arm B. Levels of HERV mRNA in bone marrow CD34+ cells and HERV specific T-cell responses at end of 1st AZA cycle and end of 6th AZA cycle (and end of treatment), respectively, in arm A vs. arm B.
Duration of azacitidine (AZA) therapy | 0-54 months
  Duration of AZA therapy in patients randomized to AZA + oral vitamin C (arm A) compared to patients randomized to AZA + placebo (arm B) assessed at end of study (EOS)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Grønbæk, Prof., MD, Study Director — Rigshospitalet, Denmark; Stine Ulrik Mikkelsen, MD, PhD, Principal Investigator — Rigshospitalet, Denmark; Ali Al-Mousawi, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (10):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev University Hospital, Copenhagen
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Goswami P, Oliva EN, Ionova T, Else R, Kell J, Fielding AK, Jennings DM, Karakantza M, Al-Ismail S, Lyness J, Collins GP, McConnell S, Langton C, Al-Obaidi MJ, Oblak M, Salek S. Paper and electronic versions of HM-PRO, a novel patient-reported outcome measure for hematology: an equivalence study. J Comp Eff Res. 2019 May;8(7):523-533. doi: 10.2217/cer-2018-0108. Epub 2019 Apr 30. PMID 31037971